CLINICAL TRIAL: NCT02067650
Title: Ultrasound Findings of Finger, Wrist and Knee Joints in Mucopolysaccharidosis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Johannes Roth, Principal Investigator, Children's Hospital of Eastern Ontario
Other Study IDs: MPSUS
Record Dates: First submitted 2013-08-13; First posted 2014-02-20 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: MPS I; MPS IV
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Hardly any imaging studies specifically addressing the articular and periarticular structures in MPS patients are available at this point. The investigators propose to do for the first time a pilot study using musculoskeletal ultrasound in patients with various types of MPS.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Mucopolysaccharidosis
* Ability to collaborate with the ultrasound assessment
* Written informed consent from parents and patients over 14 years of age, assent from children 7 to 14 years

Exclusion Criteria

* Inability to collaborate with the ultrasound assessment
* Acute trauma to a joint that will be assessed in the 3 months preceding the study
* Coexistence of other pathology that is known to affect the respective joints

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MPS I and IV
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Power Doppler | one time exam
  The primary objective is to determine whether patients with various types of MPS and at various stages of the disease exhibit abnormalities of the finger, wrist and knee joints as assessed by grey scale and Power Doppler ultrasonography.

SECONDARY OUTCOMES:
Ultrasound scanning technique | one time scan
  To determine the optimal ultrasound scanning technique for MPS patients given the potentially advanced joint contractures
Findings of synovitis or tenosynovitis | one time scan
  To determine whether there are ultrasound findings indicative of synovitis or tenosynovitis
Differences between MPS I and IV | one time scan
  To determine whether differences exist between MPS I and MPS IV
Differences between ERT and BMT | one time scan
  To determine whether differences exist between patients with or without Enzyme Replacement Therapy (ERT) or Bone Marrow Transplants
Differences between severe and attenuated phenotypes | one time scan
  To determine whether differences exist between severe and attenuated phenotypes

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Roth, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada